CLINICAL TRIAL: NCT04704479
Title: Influence of Russian Current and Expiratory Muscle Training on Expiratory Efficiency in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Russian Current and Expiratory Muscle Training in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Hassan, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002924
Record Dates: First submitted 2021-01-01; First posted 2021-01-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: expiratory muscles; dyspnea; electrical stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- combined Russian and EMT (Experimental): Russian current will be applied over the participant expiratory muscles in addition to application of EMT for more enhancement and strengthening of the expiratory muscles.
  Interventions: Device: Russian current; Device: EMT
- EMT only (Active Comparator): the participant receives EMT only over the whole study period
  Interventions: Device: EMT

INTERVENTIONS:
Device: Russian current — For application of Russian current, 2 channels with 2 electrodes each will positioned on the oblique muscles and rectus abdominis motor points using wet spongy pads to enhance electrical activity. Russian current will be a carrier frequency 2500 Hz with frequency of 5 Hz for 5 minutes of muscular conditioning, 40 Hz for 10 minutes for training of slow contraction muscular fibers and 120 Hz for 5 minutes for training of fast contraction muscular fibers with On time (contraction time) 4 secs and Off time (relaxation time) 2 secs. The contraction phase will be at time of patient's expiration while relaxation will be at time of patient's inspiration
  Other Names: NMES
  Arms: combined Russian and EMT
Device: EMT — patients in both groups trained 3 times a week, each session consisting of 1/2 h by the end of sessions. Initially, repeated cycles of 3 min of work followed by 2 min of rest were conducted (total work- time 18 min). The length of work intervals was increased on a weekly basis while rest periods were shortened to obtain a total work time of 30 min in the last week of the program. The valve opening pressure was continuously monitored at the mouthpiece to ensure the achievement of the target pressure. Patients will receive EMT with a threshold expiratory muscle trainer (Threshold; HealthScan), started breathing through the expiratory port of the threshold muscle trainer at a resistance equal to 15% of their Pemax for 1 week. The resistance will then increase incrementally, 5 to 10% each session, to reach 60% of their baseline Pemax at the end of the first month then continued at 60% of the Pemax, will be adjusted weekly to the new Pemax achieved

SUMMARY:
Respiratory muscles are essential to alveolar ventilation. In COPD, these muscles work against increased mechanical loads due to airflow limitation and geometrical changes of the thorax derived from pulmonary hyperinflation. Respiratory muscle fibers show several degrees of impairment in cellular and subcellular structures which translates, from the functional point of view, to a loss of strength (capacity to generate tension) and an increased susceptibility to failure in the face of a particular load. Expiratory Muscle Training was recommended to strengthen expiratory muscles and minimize exacerbations in addition to delaying deterioration with better functional capacity. Neuromuscular electrical stimulation (NMES) is emerging as a new rehabilitation modality for muscle strengthening that does not evoke dyspnea to obtain a benefit in patients who are unable to participate in a traditional rehabilitation program

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) remains the fourth leading cause of chronic morbidity and mortality at the global level, and it represents a major problem for public health. It is known that expiratory muscles are usually activated at the end of expiration in COPD patients during rest, or weight-bearing breathing to compensate weakness of inspiratory muscle and lung hyperinflation by time, expiratory muscle fatigue and weakness take place and more lung deterioration affecting COPD patient functional capacity occur.

The efficacy of pulmonary rehabilitation on chronic obstructive pulmonary disease (COPD) patients has been demonstrated in many studies. Although pulmonary rehabilitation is a multi-dimensional therapy, respiratory muscle training and strengthening appears to be its most effective component, expiratory muscle training improves functional exercise capacity as assessed by timed walking distance, and decreases dyspnea during daily living activities, resulting in a better health-related quality of life in patients with COPD. Russian current is a medium frequency current, which was developed for improving muscle strength. There is limited literature on the effect of Russian current in improving strength of respiratory muscles. Thus, a need arises which addresses this perspective for new management strategies

ELIGIBILITY:
Inclusion Criteria:

* Men with stage II COPD Patients
* aged from 55 to 65 years' old
* FEV1/FVC less than 70% (Patients of moderate COPD (Stage II- GOLD criteria) (Rabe et al, 2019)
* BMI 25.0-29.9 kg/m2 (Pre-obesity)
* Tobacco smokers
* No history of infections or symptom exacerbations in the previous two months before the study
* Did not participate in any selective exercise program for the respiratory muscles before

Exclusion Criteria:

* Women
* Acute exacerbation that requires a change in pharmacological management or hospitalization
* An open injury affecting the application of surface electrodes of russian current
* Asthmatic patient.
* Implanted pacemaker
* Patients with chest infection.
* Patients with pleural diseases.
* Primary valvular disease
* History of spontaneous pneumothorax
* Clinically significant peripheral vascular disease
* Severe anemia
* BMI more than 29.9 kg/m2
* Previous lung surgery
* Long-term oxygen treatment
* Patients with chronic renal failure.
* Any cognitive impairment that interferes with prescribed exercise procedures
* Musculoskeletal or neurological limitation to physical exercise
* Any patient enrolled in an anther research study for at least 30 days

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Maximum expiratory pressure | 10 weeks
  It is used to measure MEP with a pressure manometer. Measurements are usually made with patients in a sitting position and with a nose clip, Patients perform a maximal expiratory effort and sustain it for 1 to 2 seconds. The maneuver should be repeated 3 to 8 times, and the highest value recorded is used for analysis. The value obtained from the best of at least three efforts, measured at 2-min intervals, was used. Measurements will be obtained from TLC which yield higher values than those obtained of measurements from FRC

SECONDARY OUTCOMES:
dyspnea assessment | 10 weeks
  Modified Borg scale to determine degree of dyspnea and level of improvement in COPD patients. it is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during during six-minute walk testing (6MWT), 0 referred to no breathing difficulties while 10 referred to maximal difficulty of breathing
functional capacity | 10 weeks
  6 min. walking test.The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism.
COPD Assessment Test | 10 weeks
  to assess progression of lung disease, decline in functional status, and gauge effectiveness of pulmonary rehabilitation. Patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. The self-administered questionnaire consists of eight items assessing various manifestations of COPD aiming to provide a simple quantified measure of HRQoL
forced vital capacity | 10 weeks
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry. its normal value is 80% to 120%
Forced expiratory volume in the first second | 10 weeks
  Forced expiratory volume in the first second (FEV1) is the maximum amount of air that the subject can forcibly expel during the first-second following maximal inhalation. Its normal value is 80% or greater
maximal voluntary ventilation | 10 weeks
  Maximal Voluntary Ventilation (MVV) is a spirometry test that measures the largest volume that can be moved into and out of the lungs during a 10-15 second interval with voluntary effort. it reflect respiratory muscle endurance. In the normal subject MVV is about 15 to 20 times the resting minute volume.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Habib, Master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No